CLINICAL TRIAL: NCT01435837
Title: Effects of the Interaction of Caffeine and Hydration on Voice Performance
Brief Title: Interaction of Caffeine and Hydration on Voice
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Southern Illinois University Carbondale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 09433
Record Dates: First submitted 2010-09-24; First posted 2011-09-19 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Voice Disorders
Keywords: Voice; aerodynamics; acoustics
MeSH Terms: conditions — Voice Disorders | interventions — Caffeine; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeine and hydration. (Experimental): 200 mg of caffeine (over the counter caffeine tablet)
  1 liter of water
  Interventions: Drug: C2 (200mg of caffeine; 1/2 L of water); Drug: C3(200mg of caffeine; 1 L of water); Drug: C1 (200mg of caffeine, no water); Drug: Placebo (no caffeine, no water).
- No caffeine, no hydration. (Placebo Comparator)
  Interventions: Drug: C2 (200mg of caffeine; 1/2 L of water); Drug: C3(200mg of caffeine; 1 L of water); Drug: C1 (200mg of caffeine, no water); Drug: Placebo (no caffeine, no water).

INTERVENTIONS:
Drug: C2 (200mg of caffeine; 1/2 L of water) — 200mg of caffeine (tablet); 1/2 of water
  Other Names: Caffeine and water 2.
Drug: C3(200mg of caffeine; 1 L of water) — Ingestion of 200 mg of caffeine and 1 Liter of water after between pretest and posttest.
  Other Names: Caffeine and water 3.
Drug: C1 (200mg of caffeine, no water) — Ingestion of 200mg of caffeine (tablet); no water ingestion.
  Other Names: Caffeine
Drug: Placebo (no caffeine, no water). — No ingestion of caffeine; no ingestion of water between pretest and posttest.
  Other Names: Control.

SUMMARY:
The purpose of the study, Effects of Interaction of Caffeine and Hydration on Voice Performance, is to gather information about the effects of caffeine and hydration upon voice performance. The research question involves whether systemic hydration may reduce degradation on voice performance caused by caffeine ingestion. It is hypothesized that the hydration conditions will result in a less degraded vocal performance as compared with the nonhydration condition.The investigation involves abstention from any caffeine ingestion for 24 hours - from 8pm the day before testing to 8am the morning of testing. In addition, preparation for participation involves abstaining from ingesting any foods and liquids for 12 hours - from 8pm to 8am of the following morning. Each test will take about 10 minutes.

DETAILED DESCRIPTION:
The objective of this investigation is to explore the interaction of water and caffeine on voice performance through (a) acoustic measures of voice, and (b) aerodynamic measurements (minimum lung pressure required to initiate phonation. The acoustic and aerodynamic measurements were selected for this study in an effort to demonstrate the effects of four levels of hydration and caffeine status on voice quality: 1) caffeine and water1 (i.e.., Experimental Group 1 - ingestion of 200 mg of caffeine in conjunction with 500 ml of water), 2) caffeine and water2 (i.e., Experimental Group 2 - ingestion of 200 mg of caffeine in conjunction with 1.0 liter of water), 3)caffeine only (i.e., Experimental Group 3: ingestion of 200 mg of caffeine and no water), and 4) control (i.e. no ingestion of caffeine or water). The research question involves whether systemic hydration may reduce degradation on voice performance caused by caffeine ingestion. It is hypothesized that the hydration conditions will result in a less degraded vocal performance as compared with the nonhydration condition. Additionally, it is hypothesized that ingestion of 1.0 liter of water will have a greater effect on voice performance than ingestion of 500 ml of water. An additional objective of this study is to increase scientific knowledge of voice functioning by providing further data about the effect of the interaction of water and caffeine on voice performance. The results of this project may be a valuable addition to the scientific literature in vocology, and may also contribute to prevention plans for minimizing vocal disturbances. Therefore, vocational programs may include vocal prevention directions based on this study. In addition, knowledge about prevention of voice disorders may be included in the academic curriculum of students enrolled in training programs for professions involving substantial voice use.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals, ranging from 18 to 35 years of age.

Exclusion Criteria:

* History of voice disorders, history of coronary disease, history of high blood pressure.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Effect of caffeine and hydration on acoustic measures of voice. | 1 year
  The acoustic measurement of voice include the parameters of relative average perturbation (RAP), shimmer, and sound pressure level (SPL).

SECONDARY OUTCOMES:
Effect of caffeine and hydration on aerodynamic measures of voice. Effect of caffeine and hydration on aerodynamic measures of voice. | 1 year
  The aerodynamic measurement of voice includes the parameter of airflow. Airflow measurements refer to the amount of air passing through the region of the vocal folds decibels.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Claudia Franca, Ph.D., Principal Investigator — Southern Illinois University Carbondale
Locations (1):
- Southern Illinois University Carbondale, Carbondale, Illinois, United States